CLINICAL TRIAL: NCT03149562
Title: Association of Plasma Transfusions and Invasive Fungal Infection
Acronym: PT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: plasma transfusions
Record Dates: First submitted 2017-05-03; First posted 2017-05-11 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Plasma Administration; Invasive Fungal Infection; Neonatal Infection
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- plasma transfusions: The critical ill neonates with plasma transfusions
  Interventions: Drug: plasma transfusions
- non-plasma transfusions: The critical ill neonates without plasma transfusions
  Interventions: Drug: non-plasma transfusions

INTERVENTIONS:
Drug: plasma transfusions — These critical ill neonates with plasma transfusions
  Groups: plasma transfusions
Drug: non-plasma transfusions — These critical ill neonates without plasma transfusions
  Groups: non-plasma transfusions

SUMMARY:
Although lacking strong evidences, plasma transfusions are commonly used in critically ill neonates. To date, the relationships between plasma transfusions and nosocomial infection remain controversial and no study has reported the relationships between plasma transfusion and invasive fungal infection (IFI)

DETAILED DESCRIPTION:
Our aim is to explore the association between plasma transfusions and IFI in critically ill neonates

ELIGIBILITY:
Inclusion Criteria:

* all critically ill neonates admitted in hospital

Exclusion Criteria:

* severe congenital abnormality;
* died within 24 hours or left neonatal intensive care unit within 24 hours according to their parents' decisions;
* parents' decision not to participate.

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All critically ill neonates admitted in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of invasive fungal infection | 100 days
  the rate of invasive fungal infection in plasma transfusions group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China